CLINICAL TRIAL: NCT01119989
Title: Effects of a Supplementation With Amino-acids on Hepatic Lipid Metabolism
Brief Title: Effects of an Amino-acid Supplement on Hepatic Lipid Metabolism
Acronym: AMINOFRUCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: University of Bern (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: protocole 51/10
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Syndrome
Keywords: hepatic fat content; hepatic de novo lipogenesis
MeSH Terms: conditions — Metabolic Syndrome | interventions — Amino Acids; Fructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- weight maintenance diet (No Intervention)
- weight maintenance + fructose (Placebo Comparator)
  Interventions: Dietary Supplement: Fructose+maltodextrin placebo
- weight maintenance diet + fructose and amino-acid (Experimental)
  Interventions: Dietary Supplement: amino-acid + fructose

INTERVENTIONS:
Dietary Supplement: Fructose+maltodextrin placebo
  Arms: weight maintenance + fructose
Dietary Supplement: amino-acid + fructose
  Arms: weight maintenance diet + fructose and amino-acid

SUMMARY:
10 healthy male volunteers will be studied after

* a 6 day weight maintenance, balanced diet
* a 6 days weight maintenance, balanced diet supplemented with 3 grams fructose/kg body weight/day
* a 6 days weight maintenance, balanced diet supplemented with 3 grams fructose/kg body weight/day and 20g amino-acids per day At the end of each 6 days period, the following measurements will be obtained
* intrahepatic lipids (1H-MRS)
* metabolic effects of fructose ingestion (measurement of substrate oxidation, gluconeogenesis from fructose, palmitate synthesis from fructose, plasma VLDL-kinetics)

This is a randomized, double blinded study

ELIGIBILITY:
Inclusion Criteria:

* age 18-30 years
* sex: males
* BMI between 19 and 25 kg/m2
* less than 3 30min- exercise session/week

Exclusion Criteria:

* smokers
* alcohol consumption more than 50g/week
* consumption of drugs
* history of diabetes in first degree relatives
* presence of ferro-magnetic prosthesis, cardiac pacemakers, or any contra-indication to NMR

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
intrahepatic lipids | after 6 days on each controlled diet

SECONDARY OUTCOMES:
13C palmitate synthesis | after 6 days on each controlled diet

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Theytaz F, Noguchi Y, Egli L, Campos V, Buehler T, Hodson L, Patterson BW, Nishikata N, Kreis R, Mittendorfer B, Fielding B, Boesch C, Tappy L. Effects of supplementation with essential amino acids on intrahepatic lipid concentrations during fructose overfeeding in humans. Am J Clin Nutr. 2012 Nov;96(5):1008-16. doi: 10.3945/ajcn.112.035139. Epub 2012 Oct 3. PMID 23034968